CLINICAL TRIAL: NCT02118038
Title: Emotional and Cardiac Impact of Postpartum Haemorrhage. Observational Study HELP-MOM.
Brief Title: Emotional and Cardiac Impact of Postpartum Haemorrhage
Acronym: HELP-MOM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P111013; 2013-A01062-43 (Other: IDRCB)
Record Dates: First submitted 2014-03-27; First posted 2014-04-21 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Postpartum Hemorrhage Treated With Sulprostone
Keywords: Postpartum haemorrhage; Sulprostone; Cardiac impact; Emotional impact; Cardiac magnetic imaging resonance
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HELPMOM1: corresponds to the cohort of patients in whom psychological state will be studied in the immediate waning PPH then during a 6 months through appropriate questionnaires
- HELPMOM2: corresponds to the cohort of patients enrolled in group HELPMOM1 who experienced a cardiac abnormality in the initial management and will therefore be included in a cardiac monitoring

SUMMARY:
To assess the impact and to identify the main risk factors for psychological and cardiac morbidity (post-traumatic stress disorder, anxiety and depression) in case of postpartum hemorrhage

DETAILED DESCRIPTION:
The HELP- MOM study is an observational study that seeks to identify the major determinants of morbidity induced by postpartum hemorrhage (PPH) in the short and medium term. Even if PPH remains the leading cause of death in the world and in France , its main impact in so-called developed countries is not so much maternal mortality ( which is very small ) but induced morbidity.Data from the literature suggest that in a number of cases, PPH is associated with cardiac abnormalities. The nature of the abnormalities, their potential impact on the functioning of the cardiovascular system of women and their evolution over time (possibility of persistent sequelae) are not known. Similarly, it is known that the postpartum period of normal pregnancy followed by a normal delivery is at risk of psychological disorders in the mother. The PPH is a very serious situation where sometimes the vital prognosis of the mother was committed. Again, determining the exact nature and consequences of psychological harm secondary PPH are not known. Finally, fertility and the risk of recurrence after an episode PPH are also poorly understood. Outside hysterectomy hemostasis which permanently affects the fertility of the patient, the severity and type of management of PPH most likely affect fertility. Only a long-term monitoring could help address this issue. Thus, HELP MOM - study aims to address these issues. To do this, HELP MOM, was divided into two sub- studies : 1) HELP-MOM 1 "multidisciplinaire" which corresponds to the cohort of patients in whom psychological state will be studied in the immediate waning PPH then during a 6 months through appropriate questionnaires , 2 ) HELP-MOM 2 "cardio" that corresponds to the cohort of patients who experienced a cardiac abnormality in the initial management and will therefore be included in a cardiac monitoring.

ELIGIBILITY:
Inclusion Criteria:

HELPMOM1 :

* Patients with postpartum hemorrhage and receiving sulprostone
* Patient affiliated with social security

HELPMOM2 :

* Enrolled HELMOM1
* Presence of one or more items from the following list at the moment of PPH:

  * elevated troponin ("classical" or ultra) exceeds 5 times the normal value (about> 0.20 g / ml depending on the laboratory) and / or
  * electrocardiographic abnormalities (ST-segment abnormalities and / or T wave abnormalities searched in all 12 leads) and / or
  * rate of BNP (Brain Natriuretic Peptide) greater than 100 pg / m

Exclusion Criteria:

HELPMOM1:

* Age < 18 years
* Hemorrhage caused by a miscarriage, a clandestine abortion, fetal death in utero or medical or voluntary termination of pregnancy.

HELPMOM2:

- Patient with pace maker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postpartum hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Identification of risk factors for psychological impact of PPH | 1 month
  Identification of risk factors for psychological impact of PPH, as measured three questionnaires (HELPMOM1)
Occurrence of a cardiac event | Day0
  Occurrence of a cardiac event, defined as an elevation of troponin or BNP or an EKG modification during the acute phase of postpartum hemorrhage (PPH) (HELPMOM2)
Identification of risk factors for psychological impact of PPH | 3 months
  Identification of risk factors for psychological impact of PPH, as measured three questionnaires (HELPMOM1)
Identification of risk factors for psychological impact of PPH | 6 months
  Identification of risk factors for psychological impact of PPH, as measured three questionnaires (HELPMOM1)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne GAYAT, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Alexandre MEBAZAA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département Anesthésie et Réanimation - Hôpital Lariboisière, Paris, France

REFERENCES:
- [Derived] Deniau B, Ricbourg A, Weiss E, Paugam-Burtz C, Bonnet MP, Goffinet F, Mignon A, Morel O, Le Guen M, Binczak M, Carbonnel M, Michelet D, Dahmani S, Pili-Floury S, Ducloy Bouthors AS, Mebazaa A, Gayat E. Association of severe postpartum hemorrhage and development of psychological disorders: Results from the prospective and multicentre HELP MOM study. Anaesth Crit Care Pain Med. 2024 Apr;43(2):101340. doi: 10.1016/j.accpm.2023.101340. Epub 2023 Dec 19. PMID 38128731